CLINICAL TRIAL: NCT03460860
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Evaluating The Safety And Efficacy Of An Oral Supplement Containing Astaxanthin (2 mg) + Lycopene (1.8 mg) + D-Alpha-Tocopherol (10 IU) For The Treatment Of Skin Aging
Brief Title: Astaxanthin (2 mg) + Lycopene (1.8 mg) + D-Alpha-Tocopherol (10 IU) For The Treatment Of Skin Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD2017-06 (Anti-Aging Study)
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Skin Aging; Wrinkles
MeSH Terms: interventions — astaxanthine; Lycopene; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (2mg)+Lycopene (1.8mg)+D-Alpha-Tocopherol (10IU) (Experimental)
  Interventions: Dietary Supplement: Astaxanthin (2mg)+Lycopene (1.8mg)+D-Alpha-Tocopherol (10IU)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Astaxanthin (2mg)+Lycopene (1.8mg)+D-Alpha-Tocopherol (10IU) — The intervention is to be taken once daily, for 12 weeks.
  Arms: Astaxanthin (2mg)+Lycopene (1.8mg)+D-Alpha-Tocopherol (10IU)
Dietary Supplement: Placebo — The intervention is to be taken once daily, for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the clinical efficacy of a combination of Astaxanthin (2 mg), Lycopene (1.8 mg), and d-alpha-Tocopherol (10 IU) in terms of its skin anti-aging properties. Specifically, the investigators aim to determine the increase in hydration levels of the skin, decrease in atypical skin pigmentation, and reduction of signs of photoaging, particularly facial fine lines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals age 30 to 60 years old
* Fitzpatrick Skin Type I-IV
* Crow's Feet Wrinkle Scale Class 1-2
* Subjects willing to provide written informed consent

Exclusion Criteria:

* Use of topical or oral anti-aging drug therapy 1 month prior to the study
* History of allergy to cosmetics and anti-aging drugs
* History of photosensitivity reactions
* Any current or past medical condition, including seizures and stroke
* History of pigmentation disorder such as but not limited to vitiligo and leukoderma
* Immunocompromised state
* Pregnant or lactating (pregnancy kit will be used to check)
* Patients who have undergone laser, radiofrequency, peeling, and other procedural therapies for anti-aging in the month prior to the study.
* Patients with current inflammatory or infectious skin disease on the face, or history of such in the month prior to the study.
* Patients taking OCDs and other photosensitizing drugs (e.g. tetracycline).
* Not willing to provide informed consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects within each treatment group with a significant decrease in skin wrinkling measured by a validated Crow's Feet Wrinkle scale. | 12 weeks
  The scale ratings are 0 for no wrinkles, 1 for very fine wrinkles, 2 for fine wrinkles, 3 for moderate wrinkles, and 4 for severe wrinkles.

SECONDARY OUTCOMES:
Proportion of subjects within each treatment group with a significant increase in skin hydration measured by a corneometer. | 12 weeks
Proportion of subjects within each treatment group with a significant decrease in pigmentation measured by a mexameter. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- PDC Building, 1440 Taft Avenue, Manila, National Capital Region, Philippines